CLINICAL TRIAL: NCT06860971
Title: A Randomized, Double-Blind, Multicenter Phase III Clinical Trial Evaluating AL2846 Capsule Versus Placebo in Patients With Locally Advanced or Metastatic Radioiodine-Refractory Differentiated Thyroid Carcinoma Who Failed Prior VEGFR-Targeted Therapy
Brief Title: A Study of AL2846 Capsule Versus Placebo in the Treatment of Advanced Radioiodine-Refractory Differentiated Thyroid Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL2846-III-01
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AL2846 Capsules (Experimental): The treatment cycle of AL2846 Capsules is 28 days.
  Interventions: Drug: AL2846 Capsules
- AL2846 Placebo (Placebo Comparator): The treatment cycle of AL2846 Placebo is 28 days.
  Interventions: Drug: AL2846 Placebo

INTERVENTIONS:
Drug: AL2846 Capsules — AL2846 Capsule is a multi - target tyrosine kinase inhibitor, which has significant inhibitory effects on c-Mesenchymal-epithelial transition factor (c - MET), stem cell factor receptor (c - KIT), VEGFR1 and Ret Proto-Oncogene (RET).
  Arms: AL2846 Capsules
Drug: AL2846 Placebo — AL2846 Placebo without drug substance.
  Arms: AL2846 Placebo

SUMMARY:
This study aims to demonstrate that, in subjects with locally advanced or metastatic iodine - refractory differentiated thyroid cancer who have failed previous VEGFR - targeted therapy, AL2846 can significantly prolong progression - free survival (PFS) compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participants voluntarily join the study, sign the informed consent form, and demonstrate good compliance.
* Histologically or cytologically confirmed locally advanced or metastatic differentiated thyroid carcinoma (DTC).
* Age: 18 years ≤ age <75 years (calculated based on the date of signing the informed consent form).
* Eastern Cooperative Oncology Group (ECOG) performance status score: 0-1.
* Anticipated survival >12 weeks.
* At least one measurable lesion confirmed by RECIST 1.1 criteria.
* Disease progression (per RECIST 1.1) after receiving no more than 2 lines (no more than 3 types) lines of Vascular endothelial growth factor receptor tyrosine kinase inhibitor (VEGFR TKI) therapy
* Confirmed iodine-refractory status, defined by **one or more** of the following:

  1. Lesions show no iodine uptake on post-Iodine-131 therapy whole-body scan and are unlikely to benefit from further Iodine-131 therapy.
  2. Previously iodine-avid lesions progressively lose iodine uptake after Iodine-131 therapy.
  3. Mixed iodine-avid and non-iodine-avid lesions in the same patient with no biochemical response.
  4. Iodine-avid lesions with disease progression (radiologically confirmed) within 12 months.
  5. Cumulative Iodine-131 dose ≥600 mCi (22 GBq) with no disease response (radiologically confirmed).
* Thyroid stimulating hormone (TSH) ≤0.5 mIU/L under TSH-suppressive therapy.
* Laboratory parameters meeting the following criteria:

  1. Hemoglobin (HGB) ≥90 g/L.
  2. Absolute neutrophil count (NEUT) ≥1.5×10⁹/L.
  3. Platelet count (PLT) ≥90×10⁹/L.
  4. Total bilirubin (TBIL) ≤1.5×ULN.
  5. Alanine aminotransferase (ALT) and Aspartate transferase (AST) ≤2.5×ULN.
  6. Creatinine clearance (CCR) ≥50 mL/min.
  7. Prothrombin time (PT), Activated partial thromboplastin time (APTT), and International Normalized Ratio (INR) ≤1.5×ULN (without anticoagulation therapy).
  8. Serum albumin (ALB) ≥30 g/L (no albumin infusion within 7 days prior to screening).
* For participants of childbearing potential: Agreement to use effective contraception during the study and for 6 months after study completion. Females must have a negative serum/urine pregnancy test within 7 days before enrollment; males must agree to effective contraception during and for 6 months post-study.

Exclusion Criteria:

* Patients with undifferentiated thyroid carcinoma or medullary thyroid carcinoma;
* Patients who have had or currently have other malignancies. The following two situations are eligible for enrollment: other malignancies treated with a single surgery and achieving a disease - free survival (DFS) of 5 consecutive years; cured cervical carcinoma in situ, non - melanoma skin cancer, and superficial bladder tumors [Ta (non - invasive tumor), Tis (carcinoma in situ), and T1 (tumor invading the basement membrane)].
* Those with multiple factors affecting oral medications (such as difficulty in swallowing, chronic diarrhea, and intestinal obstruction, etc.);
* Adverse reactions from previous treatments have not recovered to a Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. grade score ≤ 1, except for grade 2 alopecia, grade 2 peripheral neuropathy, grade 2 anemia, non - clinically significant and asymptomatic grade 2 laboratory abnormalities, and hypothyroidism stabilized by hormone replacement therapy, and other toxicities judged by the investigator to have no safety risks.
* Known allergy to the excipient components of the study drug.
* Subjects who have participated in and used other anti - tumor clinical trial drugs within 4 weeks before randomization.
* As judged by the investigator, there are situations that seriously endanger the safety of the subject or affect the subject's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Progression - Free Survival (PFS) evaluated by the Independent Review Committee (IRC) | 34 months
  Defined as the time from the date of randomization to the date of disease progression determined by IRC or death, whichever occurred firstly.

SECONDARY OUTCOMES:
Overall Survival (OS) | 34 months
  Defined as the time from the date of randomization to the date of death for any reason.
Compare the Progression - Free Survival (PFS) evaluated by the researchers in the treatment group and the placebo group | 34 months
  PFS: The time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1.
Compare the objective response rate (ORR) between the treatment group and the placebo group | 34 months
  Objective Response Rate (ORR): It is defined as the percentage of subjects with a complete response (CR) or partial response (PR) as determined by the Independent Review Committee (IRC)/investigator according to RECIST 1.1.
Compare the Disease Control Rate (DCR) between the treatment group and the placebo group | 34 months
  Disease Control Rate (DCR): It is defined as the percentage of subjects with complete response (CR), partial response (PR), or stable disease (SD) as determined by the Independent Review Committee (IRC)/investigator according to RECIST 1.1.
Compare the Duration of Response (DOR) between the treatment group and the placebo group | 34 months
  Duration of Response (DOR): It is defined as the time from the first documented and confirmed objective response to disease progression or death from any cause (whichever occurs first), as determined by the IRC/investigator according to RECIST v1.1.
Evaluate the safety of AL2846 capsules compared with placebo in subjects with locally advanced or metastatic iodine - refractory differentiated thyroid cancer who have failed previous VEGFR - targeted therapy | 34 months
  The incidence and severity of adverse events, with severity determined according to the NCI CTCAE v5.0 grading scale.

CONTACTS AND LOCATIONS:
Locations (35):
- China (35):
  - The Second Hospital Of Anhui Medical University, Hefei, Anhui
  - cancer hospital Chinese academy of medical sciences, Beijing, Beijing Municipality
  - The Southwest Hospital of Amu, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Hospital of Guilin Medical University, Gui'lin, Guangxi
  - The Second Affiliated Hospital Of GXUST, Liuchow, Guangxi
  - The First Affiliated Hospital of Hainan Medical University, Hainan, Haikou
  - CangZhou Center Hospital, Cangzhou, Hebei
  - Harbin Medical University cancer hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of XuZhou Medical University, Xuzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - JIANGXI cancer hospital, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - JILIN cancer hospital, Changchun, Jilin
  - Liaoning Cancer Hospital, Shengyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaani
  - Xijing Hospital, Xi'an, Shaanxi
  - Shaanxi Provincial People'S Hospital, Xi'an, Shaanxi
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Weifang people's Hospital, Weifang, Shandong
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Jiaotong University School of Medicine, Tongji Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Si chuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute&Hospital, Tianjin, Tianjin Municipality
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang